CLINICAL TRIAL: NCT06650787
Title: To Study the Application of Bedside Ultrasound in Gastric Tube Placement and Determination of the Position of the End of the Gastric Tube in Children Aged 0 to 6 Years With Congenital Heart Disease
Brief Title: Application of Ultrasound Technique in Locating the End of the Gastric Tube in Children Aged 0-6 Years
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNF202333
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- According to the ultrasonic images give into stomach tube group (Experimental): According to the ultrasonic images give into stomach tube group
  Interventions: Other: Ultrasound was used to locate the end of the gastric tube
- Conventional placing nasogastric tube group (Active Comparator): Conventional placing nasogastric tube group
  Interventions: Other: Conventional placing nasogastric tube group

INTERVENTIONS:
Other: Ultrasound was used to locate the end of the gastric tube — 1. Inform the family of the purpose and method of using bedside ultrasound to guide the placement of the gastric tube, and determine the position of the end of the tube.
  2. The ultrasound machine was connected to the power supply and placed on the right side of the patient.
  3. Select the appropriate type of gastric tube and measure the length of the indwelling gastric tube by nursing staff before inserting the tube.
  4. Nurses who had been trained in ultrasound performed ultrasound judgment on the neck and abdomen of the children. Sonographers, intensive care physicians and nursing staff jointly judged the ultrasound images.
  5. Conventional judgment method was used to determine the position of gastric tube
  6. Bedside chest radiography, with results obtained by a radiologist.
  7. Keep your child safe at all times.
  Arms: According to the ultrasonic images give into stomach tube group
Other: Conventional placing nasogastric tube group — 1. Choose the appropriate type of gastric tube, and measure the length of the indwelling gastric tube by the nursing staff before the tube insertion.
  2. The gastric tube was inserted by the conventional blind insertion method.
  3. The conventional judgment method was used to determine the position of the gastric tube.
  4. Bedside chest radiography, with results obtained by a radiologist.
  5. Keep your child safe at all times.
  Arms: Conventional placing nasogastric tube group

SUMMARY:
Application of ultrasound technique to locate the end of the gastric tube in children aged 0-6 years

DETAILED DESCRIPTION:
Bedside blind insertion is the most common method for gastric tube indwelling in clinical practice. The key problem is that the position of the tube cannot be accurately determined in real time.Bedside ultrasound has become a common medical technology, and resources are easy to obtain. Therefore, bedside ultrasound has the advantages of fast, accurate, real-time repeatable, and non-invasive in determining the position of the end of the indwelling gastric tube.The purpose of this study is to investigate the accuracy of bedside ultrasound in guiding gastric tube placement and judging the position of the end of the tube in children with CHD aged 0-6 years. To explore the feasibility and effectiveness of bedside ultrasound guided gastric tube placement during perioperative period in children with congenital heart disease (CHD), this study plans to procedure the prospective randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Children with CHD who needed gastric tube in CCU were admitted
* children aged 0-6 years
* Informed consent of parents

Exclusion Criteria:

* Children with delayed sternal closure
* The parents had cognitive impairment and mental disorders

Ages: 1 Day to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of accurate gastric tube placement | The gastric tube is placed within ten minutes
  Accuracy of gastric tube placement is defined as proportion of accurate gastric tube placement (The tip of the nasogastric tube is positioned within the body or antrum of the stomach).

CONTACTS AND LOCATIONS:
Locations (1):
- CICU,Cardiovascular Center,Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China